CLINICAL TRIAL: NCT01072526
Title: Pilot Study of a Homeopathic Therapy in Combination With Cyclosporin (Restasis) in the Treatment of Dry Eye Disease
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Study personnel left institution before study completion
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LNJ-1; IRB 1095817 (Other: University of Missouri)
Record Dates: First submitted 2007-12-31; First posted 2010-02-22 (Estimated); Results first posted 2017-01-12 (Estimated); Last update posted 2017-01-12 (Estimated); Status verified 2016-11

CONDITIONS: Dry Eye Syndromes
Keywords: Dry Eye Syndromes; Lacrimal Apparatus Diseases
MeSH Terms: conditions — Dry Eye Syndromes; Lacrimal Apparatus Diseases | interventions — Lubricant Eye Drops; Cyclosporins

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Active Comparator): Subjects will receive Euphrasia-based homeopathic therapy (Artificial Tears) in combination with cyclosporin solution (Restasis) .
  Interventions: Drug: Euphrasia-based homeopathic therapy; Drug: Cyclosporin solution
- Control (Placebo Comparator): Subjects will receive placebo in combination with cyclosporin solution (Restasis) .
  Interventions: Drug: Cyclosporin solution

INTERVENTIONS:
Drug: Euphrasia-based homeopathic therapy — ophthalmic solution; 1 drop both eyes twice daily
  Other Names: Artificial Tears
  Arms: Intervention
Drug: Cyclosporin solution — Cyclosporin solution; 1 drop both eyes twice daily
  Other Names: Restasis

SUMMARY:
The purpose of this study is to determine whether a homeopathic therapy in combination with cyclosporin (Restasis) is more effective than cyclosporin (Restasis) alone in the treatment of dry eye disease.

DETAILED DESCRIPTION:
Dry eye disease affects millions of people world-wide, and presents with symptoms of blurred vision, discharge from the eyes, eye discomfort, burning, redness, sandy and gritty feeling in the eyes, and sensitivity to light. Topical eye drops for eye lubrication (i.e., artificial tear solutions) and controlling ocular inflammation through the use of topical immunomodulatory agents (i.e., cyclosporine [Restasis]) have been shown to be effective for treating dry eye syndrome, but are not curative. Recently, we have evaluated a few patients who had discontinued using Restasis as they had obtained better relief of their dry eye symptoms with a homeopathic therapy.

Potential participants will undergo an eye examination consisting of medical history and physical examination (i.e., visual acuity, pupillary exam, examination of the lids, slit-lamp examination of the conjunctiva, cornea, anterior chamber, iris, and lens, and funduscopic examination). Participants qualifying for the study will then stop all eye medications and will use a common artificial tear solution for 2 weeks prior to the baseline examination. We will evaluate 4 measures of dry eyes at baseline and after 6 weeks of therapy: 1) tear film to break-up; 2) staining of the cornea by fluorescein stain; 3) measurement of tear production over 5 minutes by Schirmer's test; and 4) the Ocular Surface Disease Index (OSDI).

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of moderate to severe dry eye syndrome with or without Sjögren's syndrome
* receiving treatment with topical cyclosporine (Restasis)
* experience one or more moderate dry eye-related symptoms, including dryness, foreign body sensation, burning, blurred vision, photophobia, and soreness or pain

Exclusion Criteria:

* history of ocular disorder including non-dry eye ocular inflammation, glaucoma, contact lens use
* trauma or surgery, including punctal plug insertion within the prior 3 months
* any uncontrolled systemic disease or significant illness
* use of topical ophthalmic medications that could affect dry eye syndrome
* pregnancy, lactation, or considering a pregnancy

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2007-12; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lenworth N Johnson, MD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri-Columbia, Mason Eye Institute, Columbia, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted Dec 2007 to Sept 2008. Participants were evaluated in the Mason Eye Institute and underwent 4 measures of dry eyes at baseline and after 6 weeks of therapy.
Pre-assignment Details: Participants will stop all common artificial tear use for 2 weeks prior to baseline examination and randomization.
Groups:
- Intervention: Euphrasia based homeopathic therapy in combination with cyclosporin (Restasis) ophthalmic solution; 1 drop both eyes twice daily. Participants to undergo 4 measures of dry eyes at baseline and after 6 weeks of therapy: 1) tear film break-up; 2) corneal staining by fluorescein; 3) Shirmer's test; and 4) Ocular Surface Disease Index (OSDI).
- Control: Cyclosporin (Restasis)ophthalmic solution; 1 drop both eyes twice daily plus placebo solution. Participants to undergo 4 measures of dry eyes at baseline and after 6 weeks of therapy: 1) tear film break-up; 2) corneal staining by fluorescein; 3) Shirmer's test; and 4) Ocular Surface Disease Index (OSDI).
Period: Overall Study
Arm/Group | Intervention | Control
Started | 6 (Study started in December 2007 (recruited 6 patients total of 20 anticipated)) | 0
Completed | 6 (Study completed in September 2008(recruited 6 patients total of 20 anticipated)) | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- 2 Arm Study - Description Below: Euphrasia based homeopathic therapy in combination with cyclosporin (Restasis)euphrasia based homeopathic therapy and cyclosporin : ophthalmic solution; 1 drop both eyes twice daily. Participants to undergo 4 measures of dry eyes at baseline and after 6 weeks of therapy: 1) tear film break-up; 2) corneal staining by fluorescein; 3) Shirmer's test; and 4) Ocular Surface Disease Index (OSDI).
Arm/Group | 2 Arm Study - Description Below
Number analyzed (Participants) | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (6.6)
Gender [Count of Participants; unit: Participants]
  Female | 4
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 6

OUTCOME MEASURES:

1. Primary Outcome: Change in Ocular Surface Disease Index (OSDI)
Description: Measures dry eye disease and effect on vision-related function. Measured on a scale of 0-100, with higher scores indicating greater disability.
Time Frame: Start of treatment, 6 weeks
Population: Any data collected was not analyzed because the study was terminated after the PI left the institution. No data is available for reporting as all study personnel have left the institution.
Groups:
- Control: cyclosporin ophthalmic solution plus placebo solution; 1 drop both eyes twice daily. Participants to undergo 4 measures of dry eyes at baseline and after 6 weeks of therapy: 1) tear film break-up; 2) corneal staining by fluorescein; 3) Shirmer's test; and 4) Ocular Surface Disease Index (OSDI).
Arm/Group | Intervention | Control
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Change in Tear Film Breakup Time
Description: Interval between last blink and break-up of tear film, measured in seconds. Less than 10 seconds = dry eye disease; lower score indicates worse disease.
Time Frame: Baseline, 6 weeks
Population: as for outcome 1
Groups:
- Control: cyclosporin (Restasis) ophthalmic solution; 1 drop both eyes twice daily. Participants to undergo 4 measures of dry eyes at baseline and after 6 weeks of therapy: 1) tear film break-up; 2) corneal staining by fluorescein; 3) Shirmer's test; and 4) Ocular Surface Disease Index (OSDI).
Arm/Group | Intervention | Control
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Change in Fluorescein Staining Scale
Description: Demonstrates abrasions on cornea and extent of disease. Graded on a scale of 0-5 with 5 being the worst score.
Time Frame: Baseline, 6 weeks
Population: as for outcome 1
Arm/Group | Intervention | Control
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Change in Schirmer Tear Test With Anesthesia Result
Description: Assesses how quickly tears are produced, measured in millimeters (mm) on blotting paper. Greater than 15 mm indicates normal tear production; lower measurement indicates presence of dry eye disease.
Time Frame: Baseline, 6 weeks
Population: as for outcome 1
Arm/Group | Intervention | Control
Number analyzed (Participants) | 0 | 0

5. Other Pre Specified Outcome: Change in Severity of Ocular Discomfort
Description: This will be calculated using a composite score of the primary and secondary outcome measures.
Time Frame: Baseline, 6 weeks
Population: as for outcome 1
Groups:
- Intervention: Subjects will receive Euphrasia-based homeopathic therapy (Artificial Tears) in combination with cyclosporin (Restasis) solution.
  Euphrasia-based homeopathic therapy: ophthalmic solution; 1 drop both eyes twice daily
  Cyclosporin solution: Ophthalmic solution; 1 drop both eyes twice daily
- Control: Subjects will receive placebo in combination with cyclosporin (Restasis) solution.
  Cyclosporin solution: Ophthalmic solution; 1 drop both eyes twice daily
Arm/Group | Intervention | Control
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | 2 Arm Study - Description Below
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 0/6

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
This study had no external sponsors. It was supported by the University of Missouri, my employer. The University of Missouri can review the data at anytime.